CLINICAL TRIAL: NCT06387979
Title: Advanced Development of Desorption Electrospray Ionization Mass Spectrometry for Intraoperative Molecular Diagnosis of Brain Cancer Using Pathology Biopsies
Status: Suspended | Type: Observational
Why Stopped: Funding issues
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 19-010725; NCI-2024-01000 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 19-010725 (Other: Mayo Clinic Institutional Review Board); R33CA240181 (NIH)
Record Dates: First submitted 2024-04-24; First posted 2024-04-29 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Glioma
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Collected samples will be stored for up to 5 years.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational: Patients undergo tissue sample collection and DESI-MS during standard of care surgery and have their medical records reviewed on study. Patients also undergo MRI per standard of care on study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-Interventional Study

SUMMARY:
This study explores whether DESI-MS can be used to identify cancerous vs. noncancerous tissue during brain tumor surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To explore the translational abilities of desorption electrospray ionization mass spectrometry (DESI-MS) as intraoperative diagnostic tool to:

Ia. Identify cancerous versus noncancerous tissue and estimate the percentage of tumor infiltration in tissue biopsies, by monitoring depletion of N-acetylaspartate (NAA) and aberrations of the phospholipid signature of neurological tissue; Ib. Identify the presence of IDH mutations by monitoring the 2-hydroxyglutarate (2HG) and therefore differentiate between IDH-mutant and wild-type gliomas.

OUTLINE: This is an observational study.

Patients undergo tissue sample collection and DESI-MS during standard of care surgery and have their medical records reviewed on study. Patients also undergo MRI per standard of care on study.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients age 18 and older
* Patients or their legally authorized representative (LAR) able to provide written consent
* Schedule to undergo tumor resection

Exclusion Criteria:

* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suspected to have glioma tumors scheduled to undergo tumor resection.
Sampling Method: Non-Probability Sample
Enrollment: 285 (Estimated)
Dates: Start 2020-10-26 (Actual); Primary Completion 2026-10-15 (Estimated); Study Completion 2026-10-15 (Estimated)

PRIMARY OUTCOMES:
Pathological state of the tissue | Up to 5 years
  Will use desorption electrospray ionization mass spectrometry (DESI-MS) to identify cancerous versus noncancerous tissue monitoring depletion of N-acetyl aspartate (NAA) and aberrations of the phospholipid signature (components of the cell membrane) of neurological tissue.
Percentage of tumor infiltration | Up to 5 years
  Will estimate the percentage of tumor infiltration in tissue biopsies by monitoring depletion of NAA and aberrations of the phospholipid signature of neurological tissue.
Presence of IDH mutations | Up to 5 years
  Will use DESI-MS to identify the presence of isocitrate dehydrogenase (IDH) mutations by monitoring the 2-hydroxyglutarate (2HG) and therefore differentiate between IDH-mutant and wild-type gliomas.

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo Quinones-Hinojosa, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

DOCUMENTS (1):
  • Informed Consent Form (2024-11-22): https://cdn.clinicaltrials.gov/large-docs/79/NCT06387979/ICF_000.pdf